CLINICAL TRIAL: NCT04694092
Title: Landiolol for Rate Control in Decompensated Heart Failure Due to Atrial Fibrillation
Acronym: LARISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Marek Sramko, Head of the Department of Acute Cardiology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LARISA2020
Record Dates: First submitted 2020-12-02; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Rapid; Acute Heart Failure; Left Ventricular Dysfunction
Keywords: rate control; betablockers; landiolol
MeSH Terms: conditions — Atrial Fibrillation; Ventricular Dysfunction, Left | interventions — landiolol

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to intensive rate control with landiolol vs. standard therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive rate control with landiolol (Experimental): Intensive heart rate control using landiolol with the goal to achieve HR<115 during the first 2 hours.
  Interventions: Drug: Intensive heart rate control with landiolol
- Standard therapy (Active Comparator): Standard heart rate control with therapy other than landiolol
  Interventions: Drug: Standard approach to heart rate control

INTERVENTIONS:
Drug: Intensive heart rate control with landiolol — Intensive heart rate control preferably with the use of short-acting betablocker landiolol in combination with digoxin
  Other Names: Rapibloc, Amomed Pharma, Austria
  Arms: Intensive rate control with landiolol
Drug: Standard approach to heart rate control — Standard heart rate control with intravenous or oral beta-blockers and/or antiarrhythmic in combination with digoxin
  Arms: Standard therapy

SUMMARY:
The study will include patients with acute heart failure with reduced left ventricular ejection fraction (<40%) triggered by atrial fibrillation (AF) with a heart rate of >130/min. Patients in cardiogenic shock, critical state, or patients requiring emergent electric cardioversion during the first 2 hours will be excluded. The patients will be randomized (1:1) to a strategy of initial intensive heart rate control using continuous infusion of landiolol and boluses of digoxin vs. standard approach to the rate control without the use of landiolol. All patients will receive recommended pharmacotherapy of acute heart failure (diuretics, nitrates, inotropes in patients with signs of low cardiac output - preferentially milrinone or levosimendan). The patients will undergo hemodynamic monitoring, laboratory testing, evaluation of symptoms, and quantification of lung water content by ultrasound for 48 hours. The study will test a hypothesis whether patients treated with initial intensive heart rate control with the preferential use of landiolol will achieve faster heart rate control, compensation of heart failure, and relief of heart failure symptoms without causing hypotension or deterioration of heart failure.

DETAILED DESCRIPTION:
Procedure:

1. Eligible patients with signed consent will be enrolled.
2. Baseline transthoracic echocardiography, laboratory testing, evaluation of subjective dyspnea, lung water by ultrasound, chest x-ray, hemodynamic monitoring (details below)
3. Randomisation 1:1 to standard therapy vs. intensive heart rate control
4. Two hours of therapy with continous hemodynamic monitoring (blood pressure by arterial line, cardiac output and stroke volume non-invasively by bioreactance)

   1. Standard therapy (oral or intravenous beta-blockers other than landiolol while avoiding hypotension or deterioration of hemodynamics, according to the preference of the physician) with a bolus of 250-500mg of digoxin
   2. Intensive heart rate control with the goal to achieve heart rate <115 during the first the hours, preferentially with continuous infusion of landiolol and a bolus of 250-500mg of digoxin. The dose will be titrated according to the actual heart rate and hemodynamic parameters (blood pressure, cardiac index, stroke volume index). If possible, in both groups, electric cardioversion will be preferentially delayed during the first 2 hours. Both groups will receive standard therapy of acute heart failure (diuretics, inotropes if needed-preferentially milrinone or levosimendan, nitrates..)
5. At 2 hours: evaluation of patients subjective dyspnea (primary clinical endpoint), heart rate (primary endpoint), hearth rhythm and hemodynamics
6. After 2 hours, both groups can be treated according to the preference of the physician.
7. Symptoms, heart rate control, hemodynamics and lung congestion will be reevaluated at 12 and 48 hours
8. The study protocol will end after 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* acute heart failure with reduced left ventricular ejection (<40%)
* atrial fibrillation with heart rate >130/min lasting presumably >12 hours and presumably contributing to the acute heart failure
* pulmonary congestion detected by auscultation, lung ultrasound or CXR

Exclusion Criteria:

* ongoing type 1. myocardial infarction
* cardiogenic shock
* presumed need for mechanical heart support during the first 48hours of the study
* presumed need for electric cardioversion during the first 2 hours of the study
* medication for heart rate control (beta-blockers, calcium channel blockers, digoxin) or antiarrhythmics introduced <24 hours before the study. Chronic therapy with these will not be a contraindication for the study
* thyreotoxicosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate control | during the first 2 hours
  Achievement of heart rate <115/min for at least 15 mins
Change in patient-reported symptoms | at 2 hours
  Change of patient-reported dyspnea evaluated 1-10 visual analog scale (1=unbearable dyspnea, 10=no symptoms)

SECONDARY OUTCOMES:
Significant change of heart rate | During the first 2 hours
  Decrease of heart rate >20% from baseline
Heart rate and heart rhythm | heart rate measured at hours 2, 12 and 48 of the study protocol
  the mean heart rate obtained from three measurements
Safety - hypotension | first 2 hours
  Occurence of hypotension requiring reduction of the dose of betablockers or vasopressors
Change in cardiac index | evaluated between baseline and hour 2
  Change in cardiac index (L/m2) evaluated noninvasively by bioreactance (Starling SV, Cheetah Medical)
Change in stroke volume index | evaluated between baseline and hour 2
  Change in stroke volume index (ml/m2) evaluated noninvasively by bioreactance (Starling SV, Cheetah Medical)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided